CLINICAL TRIAL: NCT00379743
Title: Cancer Prevention and Treatment Among African American Older Adults: Screening Trial
Brief Title: Partnership for Healthy Seniors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Centers for Medicare and Medicaid Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IRB00000063
Record Dates: First submitted 2006-09-20; First posted 2006-09-22 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Breast Cancer; Colon Cancer; Rectum Cancer; Cervix Cancer; Prostate Cancer
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Uterine Cervical Neoplasms; Prostatic Neoplasms | interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2 (Active Comparator): Individuals randomized to this arm receive the following interventions: 1) educational materials on recommended cancer-preventive services, plus 2) a health coordinator (patient navigator) who helps the participant schedule and keep appointments for cancer screening and/or treatment.
  Interventions: Behavioral: Health coordinator (or patient navigator); Behavioral: Educational materials only

INTERVENTIONS:
Behavioral: Health coordinator (or patient navigator) — Individuals randomized to receive the less intensive intervention receive educational materials only. Those randomized to the more intensive intervention are assigned a health coordinator (patient navigator) who delivers an enhanced, tailored educational intervention after review of the participant's screening history and knowledge gaps about cancer. The health coordinator also facilitate adherence to cancer screening and/or treatment services, by assisting in scheduling and keeping of appointments for cancer-related screening and/or treatment services.
Behavioral: Educational materials only — A brochure is provided to the participant with information about preventive services covered by Medicare, and the frequency with which those services should be obtained.

SUMMARY:
The Centers for Medicare and Medicaid Services (CMS) has awarded cooperative agreements to 6 sites from across the country (Salt Lake City, UT, Molokai, HI, Houston, TX, Newark, NJ, Detroit, MI, and Baltimore City) to participate in a national 4-year demonstration (September 15, 2006 to September 30, 2010). One goal of the demonstration is to reduce disparities in cancer screening among seniors from U.S. racial and ethnic minority populations. Each site will focus on a specific racial/ethnic minority group, and collaborate with CMS in project implementation. A Core questionnaire, the Cancer Screening Assessment (CSA) will be administered at baseline to all participants in the demonstration. Participant identification, randomization, and intervention implementation will be standardized across sites.

Goal: The proposal developed by the Johns Hopkins Bloomberg School of Public Health in collaboration with the Baltimore City Community Health Coalition is designed to address persistent disparities in screening for breast, cervix, colon/rectum and prostate cancer among Baltimore City's seniors.

Primary Objective: Conduct a randomized controlled trial (target N = 2,874) within a project, to compare the efficacy of 2 interventions that differ in intensity to improve continuity and outcomes of care among African Americans seniors.

Among African American seniors, compared to a less intensive intervention (general information and educational materials), does the addition of facilitation services delivered by a health coordinator result in a greater improvement in adherence to cancer screening recommendations among those who are not known to have cancer?

Study Population: We will recruit African American residents of Baltimore, age 65 years or older, and currently enrolled in Medicare Parts A and B. (Baltimore City's 82,202 seniors represent 13% of its population, and account for 68% of the City's cancer deaths. Among these seniors, 96% have Medicare Parts A and B, 54.5% have income levels at less than 250% of the federal poverty guideline, and 55.6% are African American.)

Eligible participants will respond to a baseline questionnaire, Cancer Screening Assessment (CSA). They will then be randomized to receive a less intensive or more intensive intervention. The less intensive group will receive general information about cancer and Medicare covered services, and instructions to discuss the information with their primary care doctor. The more intensive group will receive the same information as the less intensive group receives, plus tailored facilitation services delivered by a nurse-supervised community health worker. The primary outcome variable will be the difference between randomized groups in adherence to screening for breast, cervix, colon/rectum and prostate cancer.

A community advisory committee will guide all aspects of the study and will include important stake holders (both public and private sectors), representatives from the Baltimore City Community Health Coalition, the Baltimore City Department of Health, the Maryland Department of Health and Mental Hygiene, community leaders, consumers, health care providers (physicians, oncologists, nurse practitioners, physician assistants, nurses, social workers, pathologists) and academicians.

DETAILED DESCRIPTION:
Among African American seniors, compared to a less intensive intervention (general information and educational materials), does the addition of facilitation services delivered by a health coordinator result in a greater improvement in adherence to cancer screening recommendations among those who are not known to have cancer?

Background

The Centers for Medicare and Medicaid Services (CMS) received congressional authorization to launch a nationwide demonstration project to address persistent disparities in cancer prevention among racial and ethnic minority populations. Hopkins was selected as one of six national sites to conduct a demonstration project designed to test an intervention strategy to promote adherence to cancer screening among African American seniors residing in Baltimore.

Aim

This demonstration project will evaluate the efficacy of a health coordinator model in cancer screening for older African American adults in Baltimore, Maryland.

We will conduct A RANDOMIZED CONTROLLED TRIAL testing the efficacy of the model intervention in facilitating screening services for individuals who are not known to have cancer. The duration of follow-up post-randomization will be from date of randomization and September 30th, 2010, the end date for the demonstration.

We will 1) implement a population-based recruitment strategy in tandem with convenience sampling, targeting African American Medicare enrollees who reside in Baltimore, and are not known to have cancer; and 2) conduct a randomized controlled trial comparing the efficacy of a less intensive intervention (general information and educational materials in the context of "usual care") to that of a more intensive intervention, the addition of a health coordinator (HC), in promoting adherence to cancer screening.

The null hypothesis to be tested in this trial is that "the proportion of participants in the more intensive intervention group who complete at least one of the recommended screenings is equal to that of participants in the less intensive intervention group."

The primary outcome variable for the trial will be the difference between the two intervention groups in the proportion of participants who complete at least one of the recommended screenings.

Population: A total of 2874 study participants will be accrued from the Medicare enrollment database, which will be stratified by gender and age (65-74 year olds and 75 plus years).

The study population will consist of older African American Medicare beneficiaries who reside in Baltimore. The sampling frame will be restricted to African American Medicare beneficiaries, age 65 and older, Baltimore residents enrolled in Medicare Parts A and B, but not enrolled in managed care (Medicare Part C), hospice, or some other extended care facility. With a population of 651,154, African Americans constitute 64% of Baltimore City's total population44. Additionally, 13.2% of Baltimoreans are age 65 or older, and this accounts for 68% of the City's cancer deaths.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or older;
* Residence in Baltimore;
* Enrolled in Medicare Part A;
* Enrolled in Medicare Part B of Title XVIII of the Social Security Act;
* Provided informed consent;
* Must be free from cancer or in remission for 5 years or more

Exclusion Criteria:

* Age less than 65;
* Residence outside of Baltimore;
* Enrollment in Medicare managed care (Part C);
* Residence in a chronic care facility or otherwise institutionalized;
* Planning to move within the next year;
* Unable or unwilling to give informed consent;
* Diagnosed with cancer within 5 years or less;
* Diagnosed with cancer more than 5 years ago, but cancer in remission for less than 5 years

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 2593 (Actual)
Dates: Start 2006-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Difference between the two intervention groups in the proportion of participants who complete at least one of the recommended screenings. | Number of days from date of randomization to date of completion of participation in the study

SECONDARY OUTCOMES:
Adherence to maintenance screening. | Number of days beyond extended window for completion of a specific screening test
Timely notification of abnormal screening results. | Number of days between detection of an abnormal screening result and participant notification about the results
Timely follow up with specialist following abnormal screening result. | From date of detection of an abnormal screening result to date of visit with specialist
Timely diagnosis following abnormal result. | From date of detection of an abnormal screening result to date of diagnosis
Timely treatment start-up. | Number of days from the date of diagnosis to date of initiation of therapy
Improved utilization of Medicare-covered preventive services. | From date of randomization to date of completion of participation in the study
Stage at diagnosis. | At the time of diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Dobs, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Bloomberg School of Public Health, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Martinez KA, Pollack CE, Phelan DF, Markakis D, Bone L, Shapiro G, Wenzel J, Howerton M, Johnson L, Garza MA, Ford JG. Gender differences in correlates of colorectal cancer screening among Black Medicare beneficiaries in Baltimore. Cancer Epidemiol Biomarkers Prev. 2013 Jun;22(6):1037-42. doi: 10.1158/1055-9965.EPI-12-1215. Epub 2013 Apr 29. PMID 23629519